CLINICAL TRIAL: NCT06705777
Title: Self-Paired Clinical Study of the Combination of Aesculus Hippocastanum 10 mg, Polygonum Acre 10 mg, Smilax Papyracea 40 mg, Rutin 20 mg Tablets in Grade 1, 2 or 3 Hemorrhoidal Disease After 60 Days of Treatment
Brief Title: Randomized Study of Oral Aesculus Hippocastanum and Combinations in Hemorrhoidal Disease After 60 Days of Treatment
Acronym: RSFAhCHD60T
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other); Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Carlos Pereira Nunes, Professor, Fundação Educacional Serra dos Órgãos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7.078.287; 83102224.6.0000.5247 (Other: Certificado de Apresentação de Apreciação Ética - Anvisa)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Haemorrhoidal Disease
MeSH Terms: interventions — horse chestnut seed; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aesculus hippocastanum, and interventions (Other): Self-paired study
  Interventions: Drug: Aesculus hippocastanum, and interventions

INTERVENTIONS:
Drug: Aesculus hippocastanum, and interventions — venotonic
  Other Names: Vastonic

SUMMARY:
To demonstrate the clinical efficacy of the combination of Aesculus hippocastanum, Polygonum acre, Smilax Pepyracea, and rutin in tablets in improving local symptoms (bleeding, pain, thrombosis, perianal dermatitis, hemorrhoidal nipple prolapse) assessed using a 100mm visual scale (VAS) over 60 days among adult patients with grade 1, 2 or 3 hemorrhoidal disease.

DETAILED DESCRIPTION:
Hemorrhoidal disease (HD) is the most common proctological condition, with an up to 86% prevalence (asymptomatic individuals underestimated). It is expected that 5% of the population might have at least one episode of HD during their lifetime, most individuals amenable to medical therapy but 10 to 20% of them requiring surgical intervention. HD has an occurrence peak between the 5th and 7th decades of life. Haemorrhoids can be defined as varicose dilatation of the submucosal anorectal veins due to persistently elevated venous pressure in the hemorrhoidal plexus, that is, they develop when the venous drainage of the anus and rectum is altered, causing dilatation of the venous plexus and connective tissue, creating an overgrowth of the anal mucosa of the rectal wall. The term HD is used when haemorrhoids cause symptoms. Aesculus hippocastanum (horse chestnut), rutin, Smilax papyracea (sarsaparilla), Polygonum acre (dotted smartweed) combination is commonly used to control chronic venous insufficiency (CVI) manifestations. Assuming pathophysiology of HD and CVI are similar, the investigators hypothesized the above combination could be also useful in the management of the former condition.

ELIGIBILITY:
Inclusion Criteria:

* Grade 1, 2 or 3 hemorrhoidal disease
* Complaints related to haemorrhoidal disease/acute hemorrhoidal crisis (defined as acute anal pain due to haemorrhoidal prolapse with or without bleeding, edema and thrombosis)
* For female patients of reproductive age, not pregnant or breastfeeding, using reliable contraception.
* Patient has read, understood, signed and dated the informed consent form

Exclusion Criteria:

* Presence of concomitant severe systemic disorders
* Treatment with venotonics within 2 months of the date of inclusion in the study
* Women of reproductive age who are pregnant or breastfeeding, or who do not wish to use contraception during the study period.
* Known allergy or hypersensitivity to any component of the study medication
* Known significant laboratory abnormality
* Anal fissure
* Inflammatory bowel disease
* Colorectal cancer
* Anal abscess or fistula
* Previous anorectal surgery and/or radiotherapy in the pelvic-perineal region
* Patient with a change in general condition that is incompatible with her participation in the study
* Patient who wishes to become pregnant within 6 months
* Inability of the patient to understand the nature of the study and follow the doctor's recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-22 (Actual)

PRIMARY OUTCOMES:
Hemorrhoidal Disease Symptom Score (HDSS) (adapted) | 2 months
  4 questions:
  1. How often do you feel pain because of your hemorrhoids?
  2. How often do you experience itching or discomfort in your anus?
  3. How often do you bleed when you have a bowel movement?
  4. How often do you soil your underwear (anal soil)?
  Possible answers:
  * Never
  * Less than once a month
  * Less than once a week
  * 1 to 6 days a week
  * Every day (always)
Short Health Scale HD (SHSHD) | 2 months
  1. In your opinion, how severe are your symptoms caused by hemorrhoids?
  2. Do your symptoms interfere with your daily activities?
  3. Are your symptoms causing you a lot of concern?
  4. How is your overall sense of well-being?
  Possible answers:
  * 1
  * 2
  * 3
  * 4
  * 5

SECONDARY OUTCOMES:
global satisfaction of the patient | 3 months
  Please indicate your overall satisfaction with the effectiveness of your treatment to date on the scale below:
  * Bad
  * Acceptable
  * Good
  * Very Good
global satisfaction of the physician | 3 months
  Please indicate your overall satisfaction with the effectiveness of your treatment to date on the scale below:
  * Bad
  * Acceptable
  * Good
  * Very Good

OTHER OUTCOMES:
Effectiveness in hemorrhoidal symptoms | 3 months
  The 100mm visual scale is assessed by the patient between "0" = absence of venous symptoms and "100" = maximum intensity of symptoms. The visual scale is performed by the patient in the presence of the investigator. This visual scale assesses the symptoms of haemorrhoidal disease in a global manner: bleeding, pain, thrombosis, perianal dermatitis (pruritus or anal discomfort), prolapse of the hemorrhoidal nipple, soiling.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Nunes, Professor, Principal Investigator — Fundação Educacional Serra dos Órgãos
Locations (1):
- Centro Universitário Serra dos Órgãos - UNIFESO, Teresópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acheson AG, Scholefield JH. Management of haemorrhoids. BMJ. 2008 Feb 16;336(7640):380-3. doi: 10.1136/bmj.39465.674745.80. No abstract available. PMID 18276714
- [Background] Ba-bai-ke-re MM, Huang HG, Re WN, Fan K, Chu H, Ai EH, Li-Mu MM, Wang YR, Wen H. How we can improve patients' comfort after Milligan-Morgan open haemorrhoidectomy. World J Gastroenterol. 2011 Mar 21;17(11):1448-56. doi: 10.3748/wjg.v17.i11.1448. PMID 21472103
- [Background] Bartolo M. [Socioeconomic impact of venous diseases in Italy]. Phlebologie. 1992 Nov-Dec;45(4):423-31. French. PMID 1302317
- [Background] Bergan JJ, Schmid-Schonbein GW, Coleridge Smith PD, Nicolaides AN, Boisseau MR, Eklof B. Chronic venous disease. Minerva Cardioangiol. 2007 Aug;55(4):459-76. No abstract available. English, Italian. PMID 17653022
- [Background] Belczak SQ, Sincos IR, Campos W, Beserra J, Nering G, Aun R. Veno-active drugs for chronic venous disease: A randomized, double-blind, placebo-controlled parallel-design trial. Phlebology. 2014 Aug;29(7):454-60. doi: 10.1177/0268355513489550. Epub 2013 May 16. PMID 23761871
- [Background] Zagriadskii EA, Bogomazov AM, Golovko EB. Conservative Treatment of Hemorrhoids: Results of an Observational Multicenter Study. Adv Ther. 2018 Nov;35(11):1979-1992. doi: 10.1007/s12325-018-0794-x. Epub 2018 Oct 1. PMID 30276625
- [Result] Dickson S, Gallagher J, McIntyre L, Suter A, Tan J. An open study to assess the safety and efficacy of Aesculus hippocastanum tablets (Aesculaforce 50mg) in the treatment of chronic venous insufficiency. J Herb Pharmacother. 2004;4(2):19-32. PMID 15364642
- [Result] Park G, Kim TM, Kim JH, Oh MS. Antioxidant effects of the sarsaparilla via scavenging of reactive oxygen species and induction of antioxidant enzymes in human dermal fibroblasts. Environ Toxicol Pharmacol. 2014 Jul;38(1):305-15. doi: 10.1016/j.etap.2014.06.009. Epub 2014 Jun 28. PMID 25022355
- [Result] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751
- [Result] Perera N, Liolitsa D, Iype S, Croxford A, Yassin M, Lang P, Ukaegbu O, van Issum C. Phlebotonics for haemorrhoids. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD004322. doi: 10.1002/14651858.CD004322.pub3. PMID 22895941